CLINICAL TRIAL: NCT02898519
Title: Serological Response in Patients Infected by Leptospirosis 1 to 7 Years Earlier
Brief Title: Immune Response After Leptospirosis Infection
Acronym: SERO7LEPTO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 2015/CHU/07
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Leptospirosis
MeSH Terms: conditions — Leptospirosis | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cohort — Blood sampling

SUMMARY:
Leptospirosis is a zoonotic infection induced by pathogen bacteria (genus: Leptospira) growing in water polluted by animal fluids. Due to its 10 fold occurence in French overseas aera, and especially in Reunion Island, as compared to metropoly, it is considered as a major public health issue.

An important inter-individual variability in humoral immune response suggests that vaccination should be recommended in exposed subjects.

This cohort study aimed to determine if subjects that have been infected by leptospirosis for 1 to 7 years still remain immunized, and then do not need vaccination.

DETAILED DESCRIPTION:
Every year more than 500 000 severe forms of leptospirosis are diagnosed in Reunion Island. The risk of mucocutaneous contact with contaminated media remains important due to highly aqueous environment.

Cured subjects that have been infected for 1, 2, 3, 4, 5, 6 or 7 years will be enrolled. The qualitative and quantitative humoral immune response to leptospirosis infection will also be evaluated to determine whether they still get protective immunization. Leptospirosis immunization will be evaluated using micro-agglutination test.

Graded immune responses related to the severity and the length of the infection will also be investigated.

Finally, 3 methods used for leptospirosis diagnosis will be compared. It is expected from this study to evaluate the appropriate conditions in which new vaccination could be required to prevent further leptospirosis infection in cured subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed for leptospirosis by polymerase chain reaction measured in Reunion Island Hospital between 209-2015
* with social security issue

Exclusion Criteria:

* Leptospirosis diagnosis not confirmed by polymerase chain reaction
* subject exhibiting immunodepressive status (cancers, transplantation, immune deficit, blood disorders)
* under medication: corticoids, immunosuppressor, chemiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Leptospirosis-cured subjects that have undergone leptospirosis
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Leptospirosis immunization assessed by serum immunoglobulin | 1-7 years after leptospirosis infection
  Humoral immune response will be measured in serum cured-subjects using micro-agglutination test

SECONDARY OUTCOMES:
rate of still-immunized patients | 1-7 years after leptospirosis infection
  Seropositive subjects will be measured using the ELISA serion method and the ELISA recombinant protein method
comparison of 3 diagnosis method for leptospirosis | 1-7 years after leptospirosis infection
  Matched results of the 3 methods: micro-agglutination test, ELISA serion method and ELISA recombinant protein method will be compared

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS TRAVERSIER, MD, Principal Investigator — CHU DE LA REUNION

IPD SHARING:
Plan to Share IPD: No